CLINICAL TRIAL: NCT00840580
Title: Prospective, Randomized Study Comparing Effect on Wound Healing of Vigamox (Moxifloxacin 0.5% Ophthalmic Solution) and Cravit (Levofloxacin 0.5% Ophthalmic Solution) Administered Post-Surgically in Patients Undergoing Cataract Extraction
Brief Title: Effect on Wound Healing of Vigamox Versus Cravit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMA-08-22
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Cataract Extraction
Keywords: Cataract, Cornea, Vigamox, Cravit
MeSH Terms: conditions — Cataract; Corneal Diseases | interventions — Moxifloxacin; Ophthalmic Solutions; Levofloxacin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vigamox (Experimental): One drop 4 times a day in study eye for one week prior to surgery, followed by one drop 4 times a day for two weeks beginning Day 1 post surgery.
  Interventions: Drug: Moxifloxacin 0.5% ophthalmic solution (Vigamox)
- Cravit (Active Comparator): One drop 4 times a day in study eye for one week prior to surgery, followed by one drop 4 times a day for two weeks beginning Day 1 post surgery.
  Interventions: Drug: Levofloxacin 0.5% ophthalmic solution (Cravit)

INTERVENTIONS:
Drug: Moxifloxacin 0.5% ophthalmic solution (Vigamox) — One drop 4 times a day in study eye for one week prior to surgery, followed by one drop 4 times a day for two weeks beginning Day 1 post surgery.
  Other Names: Vigamox
  Arms: Vigamox
Drug: Levofloxacin 0.5% ophthalmic solution (Cravit) — One drop 4 times a day in study eye for one week prior to surgery, followed by one drop 4 times a day for two weeks beginning Day 1 post surgery.
  Other Names: Cravit
  Arms: Cravit

SUMMARY:
The purpose of this study was to compare the effects of Vigamox and Cravit on corneal wound healing after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any race and either sex, and over the age of 18, who are scheduled for removal of a cataract and implantation of a posterior chamber intraocular lens using clear corneal incisions or near-clear corneal incisions.
* Intraocular pressure (IOP) readings, treated or untreated, less than or equal to 20 mmHg prior to surgery. Glaucoma patients are eligible if an ocular hypotensive agent (only one) controls their IOP.
* Other than cataracts, have normal healthy eyes as determined by the ophthalmic examination and case history.
* Subconjunctival injections right after cataract surgery are allowed.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any cataract wound that is stitched or any gross abrasion of the epithelium after removal of a cataract and implantation of a posterior chamber intraocular lens.
* Fluorescein staining of the cornea at baseline.
* History or evidence of ocular or systemic disease, which would preclude participation in this study. Examples could include autoimmune disease affecting the cornea as well as any corneal dystrophies.
* History of ocular inflammatory disease, ocular herpes infection, iritis, uveitis, or Sjögren's syndrome.
* Known or suspected allergy or hypersensitivity to levofloxacin or any related medicines, such as cinoxacin (Cinobac), ciprofloxacin (Cipro or Ciloxan), norfloxacin (Chibroxin or Noroxin), ofloxacin (Floxin), or nalidixic acid (NegGram), preservatives, dyes, or any components of the study medication.
* Treatment for an ocular infection within 30 days prior to study entry.
* Use of topical or systemic steroids within 7 days prior to study entry.
* Use of topical anti inflammatory drugs within 7 days prior to study entry.
* Pregnancy, nursing/lactation, or inadequate birth control methods. Oral contraceptives are allowed.
* Patients with uncontrolled diabetes and/or diabetic retinopathy.
* No ointment is used after cataract surgery.
* Other protocol-defined exclusion criteria may apply.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with epithelial defect | Day 1, Day 2, Day 3, Day 10
  The eye was imaged. An epithelial defect was defined as a non-continuous epithelium. The eye was considered healed when the defect was no longer visible.

CONTACTS AND LOCATIONS:
Overall Officials: Eung Kweon Kim, MD/PhD, Principal Investigator — Severance Hospital, Yousei University College of Medicine
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Derived] Han KE, Chung WS, Kim TI, Kim S, Kim T, Kim EK. Epithelial wound healing after cataract surgery comparing two different topical fluoroquinolones. Yonsei Med J. 2014 Jan;55(1):197-202. doi: 10.3349/ymj.2014.55.1.197. PMID 24339307